CLINICAL TRIAL: NCT05043870
Title: Combination Therapy of Infliximab and Immunosuppressives for Pediatric Crohn's Disease
Brief Title: Combined Immunosuppression for Pediatric Crohn's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Head of department of gastroenterology, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combined therapy in CD
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease; Infliximab; Immunosuppression; Children, Only
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Immunosuppressive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- infliximab and immunosuppressives therapy (Experimental): the infusion of infliximab (IFX) (5mg/kg) were given at 0, 2, 6 weeks and then every 8 weeks, the immunomodulatory agent was azathioprine 1-2mg/kg per day or methotrexate 10-25 mg/m2 week
  Interventions: Drug: Infliximab and immunosuppressives
- infliximab therapy (Active Comparator): the infusion of infliximab (IFX) (5mg/kg) were given at 0, 2, 6 weeks and then every 8 weeks
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab and immunosuppressives — the infusion of IFX (5mg/kg) were given at 0, 2, 6 weeks and then every 8 weeks, the immunomodulatory agent was azathioprine 1-2mg/kg per day or methotrexate 10-25 mg/m2 week
  Other Names: IFX, IMMs, AZA, MTX
  Arms: infliximab and immunosuppressives therapy
Drug: Infliximab — the infusion of IFX (5mg/kg) were given at 0, 2, 6 weeks and then every 8 weeks
  Other Names: IFX
  Arms: infliximab therapy

SUMMARY:
This is a randomized controlled trial to compare the efficacy and safety of infliximab and immunosuppressives therapy alone or in combination for pediatric Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. 6-18 years old
2. diagnosis of Crohn's Disease
3. Pediatric Crohn's disease Activity Index (PCDAI)>30 or The Simple Endoscopic Score for Crohn Disease (SES-CD) >10 before treatment
4. receiving exclusive enteral nutrition or corticosteroids as first-line treatment, Pediatric Crohn's disease Activity Index (PCDAI)>10 or The Simple Endoscopic Score for Crohn Disease (SES-CD)≥3 after exclusive enteral nutrition or corticosteroids
5. The patient or legal guardian sign the informed consent documents

Exclusion Criteria:

1. history of biological agents targeting at tumor necrosis factor (TNF)
2. Crohn's Disease-related surgery
3. infections
4. tumors

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical remission | week 54
  The clinical remission rate at week 54
endoscopic remission | week 54
  The endoscopic remission rate at week 54

SECONDARY OUTCOMES:
Pediatric Crohn's disease Activity Index score | week0, week2, week6, week14, week22, week30, week38, week46, week54
  The Pediatric Crohn's disease Activity Index (PCDAI) was assessed at each infusion point. PCDAI score ranges from 0 to 100, the higher means the worse outcome.

OTHER OUTCOMES:
infliximab concentration | week 14, 38
  The infliximab (IFX) concentration and anti-infliximab antibodies (ATI) were measured before the infusion of week 14, 38.
adverse events | within one year
  The rate of the potential adverse events were monitored during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China